CLINICAL TRIAL: NCT04507854
Title: Return to Performance Criteria Following Shoulder Instability Surgery in the Athlete.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Principal Investigator, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 04082020
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Shoulder; Return to Sport; Surgery
MeSH Terms: interventions — Range of Motion, Articular; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operated athletes (Experimental)
  Interventions: Other: Strength, range of motion and functional tests + Questionnaire

INTERVENTIONS:
Other: Strength, range of motion and functional tests + Questionnaire — Patients undergoing instability surgery will perform amplitude, strength, functional tests and a questionnaire at 6 months of the operation. Then they will be contacted at 12, 18 and 24 months to find out if they have regained their performance level or if they have injured their shoulder again.

SUMMARY:
The purpose of this study is to determine whether certain criteria for returning to the field can be predictive of a return of the athlete to a level of performance similar to that of before his shoulder injury. In this context, these different criteria will be tested at 6 months in post-surgery while performance monitoring will be carried out at 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Athletes playing sports soliciting the upper limb (> 3 hours per week)
* Athletes between 18 and 35 years of age
* Patients with recent Bankart or Latarjet shoulder surgery (less than 4 months ago)
* Patients accepting the study protocol

Exclusion Criteria:

* Patients with other pathologies that interfere with planned physical activity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Strength test | 6 months from the surgery
  The strength will be assess with a isokinetic device. It will allow to calculate the maximum force of the subject at the level of the rotators of the shoulder. This is a dorsal decubitus test. The subject's arm will be positioned in 90° of abduction of shoulder abduction.
  In this position, the subject will perform tests at different speeds (60°/s concentric, 240°/s concentric and 60°/s eccentric). This will calculate the maximum force.
Range of motion | 6 months from the surgery
  This test will consist of a measurement of the active and passive joint amplitudes of the athlete.
  Different movements will be tested:
  flexion, extension, abduction, external rotation elbow to body, hand-back, internal/external rotations at 90° arm abduction in frontal plane.
Functional test | 6 months from the surgery
  Two functional tests will be proposed, one closed chain and the other open chain. Athletes will realize the one that comes closest to their daily practice.
  The Upper Quarter Y-Balance test will be performed by athletes in closed-chain sports.
  The second proposed test will be the medicine ball throw.
Questionnaire DASH | 6 months from the surgery
  The questionnaire that athletes will complete will be the DASH (Disabilities of the Arm, Shoulder and Hand Scale) questionnaire.
Follow-up questionnaire at 12 months | At 12 months from the surgery
  Athletes will be asked to answer different questions about their performance level since their sports restart at 12, 18 and 24 months post-operation.
  We will also look into a possible recurrence of injury to their shoulder.
Follow-up questionnaire at 18 months | At 18 months from the surgery
  Athletes will be asked to answer different questions about their performance level since their sports restart at 12, 18 and 24 months post-operation.
  We will also look into a possible recurrence of injury to their shoulder.
Follow-up questionnaire at 24 months | At 24 months from the surgery
  Athletes will be asked to answer different questions about their performance level since their sports restart at 12, 18 and 24 months post-operation.
  We will also look into a possible recurrence of injury to their shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Belgium